CLINICAL TRIAL: NCT01102062
Title: Human Urinary Biomarker for Orange Juice Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 557-ICL-649
Record Dates: First submitted 2010-04-07; First posted 2010-04-12 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orange Juice (Experimental): 1 glass (=200mL) of orange juice
  Interventions: Dietary Supplement: orange juice

INTERVENTIONS:
Dietary Supplement: orange juice

SUMMARY:
Human urinary metabolic profiling showed to be very successful to elucidate biomarkers linked to geographic origin and specific food consumption patterns (Holmes and Loo et al.: Human metabolic phenotype diversity and its association with diet and blood pressure. Nature 2008:1-6). It was possible to identify urinary metabolites directly linked to animal vs. vegetable protein intake. This is very valuable for future population studies, where diet is an important lifestyle factor but food questionnaires are time-consuming and expensive. Moreover, miss-reporting is a very common problem.

Our hypothesis is to find the same biochemical marker for orange juice as we already found in a preceding nutritional studies where participants recorded orange consumption.

DETAILED DESCRIPTION:
To elucidate the citrus fruit biomarker it needs to be ensured that all volunteers do not consume citrus fruits and foods potentially containing similar ingredients. Therefore it is necessary to ask volunteers to refrain from these foods by giving them dietary restrictions. Extensive literature research showed that some foods (such as grain legumes and brie cheese) may contain the same compound, but in much smaller amounts.

Days 1-3 will be on open diet but with dietary restrictions (no alcohol, cheese, fruits, ethnic foods such as Chinese and Indian food, grain legumes such as beans, lentils, peas and peanuts, and all kinds of sprouts (such as cress or alfalfa)). On day 2 a glass of orange juice (200ml) will be consumed in addition to the open diet. Urine collection will continue and stop on day 4 at 10 am.

During the study to minimise variation in biomarker excretion due to other beverages the participants beverage intake will be restricted to water and coffee.

All urine samples will then be analysed using high resolution NMR spectroscopy and mass spectrometry. Mathematical data analyses as well as the visual examinations of the NMR spectra will also be carried out to validate the presence of citrus fruit biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* male/female
* aged 18-45 years
* non-smoker
* BMI 18-25 kg/m2

Exclusion Criteria:

* regular drug intake
* regular food supplements intake

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To elucidate urinary biochemical markers for the consumption of orange juice. | 6 months
  1H NMR urinary metabolite spectra will be acquired. Proline betaine will be quantified by peak integration of the resonance at 3.11ppm in the NMR spectrum.

SECONDARY OUTCOMES:
To investigate the kinetics of elucidated biomarker excretion over time. | 6 months
  Excretion of proline betaine, as quantified from the 1H NMR spectrum of urine, will be plotted over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Heinzmann SS, Brown IJ, Chan Q, Bictash M, Dumas ME, Kochhar S, Stamler J, Holmes E, Elliott P, Nicholson JK. Metabolic profiling strategy for discovery of nutritional biomarkers: proline betaine as a marker of citrus consumption. Am J Clin Nutr. 2010 Aug;92(2):436-43. doi: 10.3945/ajcn.2010.29672. Epub 2010 Jun 23. PMID 20573794